CLINICAL TRIAL: NCT04971577
Title: Efficacy of Simvastatin in Reducing Liver Fibrosis in Patients With Advanced Fibrosis Due to Alcohol: Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy of Simvastatin in Alcoholic Liver Fibrosis
Acronym: SIMFIB
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Project manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIMFIB
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Liver Fibrosis; Alcohol Abuse
MeSH Terms: conditions — Liver Cirrhosis; Alcoholism | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Placebo Comparator)
  Interventions: Drug: Simvastatin 40mg
- Treatment arm (Experimental)
  Interventions: Drug: Simvastatin 40mg

INTERVENTIONS:
Drug: Simvastatin 40mg — participants will receive a capsule containing 4 tablets simvastatin 10 mg (40 mg total) every 24 hours at night

SUMMARY:
Evaluate the efficacy of simvastatin in reducing liver fibrosis in patients with advanced fibrosis due to alcohol

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Chronic alcohol-related liver disease according to international guidelines (EASL, European Association for the Study of the Liver) and with data of significant liver fibrosis obtained in the diagnostic biopsy at the beginning of the study or in the last biopsy of the patient within 6 months prior to randomization. Significant liver fibrosis is defined by a score on the Ishak fibrosis scale of between 3 and 6.
3. Patients in the compensated chronic liver disease phase defined by the absence of clinical decompensations at the time of entering the study, with or without data of portal hypertension.
4. Women of childbearing potential must have a negative urine pregnancy test prior to study enrollment and agree to use highly effective contraceptive methods (combined oral pill, injectable or implanted contraceptive, intrauterine device / hormone delivery system intrauterine) during the study.

Exclusion Criteria:

1. Patients receiving statins or fibrates.
2. Patients with other etiologies of liver disease in addition to alcohol: hepatitis C, hepatitis B, autoimmune hepatitis, Wilson's disease, or hemochromatosis.
3. Patients in whom hepatitis C has been cured with antivirals in the 2 years prior to inclusion in the study.
4. Patients with a CK elevation of 50% or more above the upper limit of normal at the time of study inclusion.
5. Gastrointestinal bleeding due to portal hypertension within 12 months prior to inclusion in the study.
6. Clinical hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy, in the 12 months prior to inclusion in the study.
7. Patients in need of diuretic treatment in the previous 12 months to control ascites or hydrothorax.
8. Spontaneous bacterial peritonitis within 12 months prior to study enrollment.
9. Hepatocellular carcinoma of any stage.
10. Patients with known muscle disease.
11. Patients with previous rhabdomyolysis.
12. Patients being treated with strong CYP3A4 enzyme inhibitors (see section 5.2: Concomitant drugs, not allowed and allowed).
13. Patients being treated with drugs with possible interactions with simvastatin (see section 5.2: Concomitant drugs, not allowed and allowed).
14. Patients with a history of significant extrahepatic disease with poor short-term prognosis, including New York Heart Association Grade III / V congestive heart failure, GOLD COPD> 2, chronic kidney disease with serum creatinine> 2mg / dL or under therapy of kidney replacement.
15. Patients with extrahepatic malignancies, including solid tumors and hematologic malignancies.
16. Patients with a history or increased risk of intestinal obstruction.
17. Pregnancy or breastfeeding.
18. Patients included in other clinical trials during the previous month.
19. Patients with mental disabilities, language barriers, poor social support or any other reason considered by the researcher as essential for adequate understanding, cooperation or compliance with the study.
20. Presence of data on alcoholic hepatitis in liver biopsy upon inclusion.
21. Patients with contraindications for statins.
22. Known hypersensitivity to simvastatin.
23. Refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline biopsy in histological fibrosis Ishak score (0-4 range. higher scores mean a worse result) | 18 months
  Change from range baseline biopsy in histological fibrosis score measured through the Ishak scale at 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Gines, Md, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Jordi Gratacos, Barcelona, Spain

REFERENCES:
- [Derived] Luo X, Wang G, Yang L, Hernandez-Gea V. Future research direction of portal hypertension based on Baveno VII. Chin Med J (Engl). 2025 Sep 20;138(18):2268-2282. doi: 10.1097/CM9.0000000000003785. Epub 2025 Aug 18. PMID 40824526